CLINICAL TRIAL: NCT01060137
Title: Evaluation of the Usefulness of DurogesicD-TRANS for Pain Treatment in Lung Cancer Patients
Brief Title: Fentanyl Matrix in Lung Cancer Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: R&D Director, Janssen Korea, Ltd., Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR012259
Record Dates: First submitted 2010-01-29; First posted 2010-02-02 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2010-02

CONDITIONS: Lung Cancer; Pain
Keywords: fentanyl matrix
MeSH Terms: conditions — Lung Neoplasms; Pain

ARMS (1):
- 001 (Experimental): fentanyl matrix Fentanyl transdermal patch 12 - 25mcg/hr can increase with 12 - 25mcg/h based on pain assessment
  Interventions: Drug: fentanyl matrix

INTERVENTIONS:
Drug: fentanyl matrix — Fentanyl transdermal patch 12 - 25mcg/hr

SUMMARY:
The purpose of this study is to evaluate the usefulness of fentanyl matrix by assessing patients' satisfaction when administrating fentanyl matrix, a background pain treatment, and a breakthrough pain treatment to lung cancer patients who complain of pain. Fentanyl matrix is designed to deliver medication at a nearly constant amount per unit time into the body through the skin for 3 days (72 hours).

DETAILED DESCRIPTION:
This study is open-label, single-arm, multicenter, prospective study to evaluate the usefulness of fentanyl matrix (fentanyl transdermal patch-type system) by assessing patient satisfaction when administrating fentanyl matrix (a background pain treatment, and a breakthrough pain treatment) for patients with lung cancer for 21 days. Fentanyl transdermal patch-type system is designed to deliver medication at a nearly constant amount per unit time into the body through the skin for 3 days (72 hours). Studies about transdermal fentanyl have found that it had analgesic effects on malignant pain, and most patients receiving the medication preferred fentanyl because they experienced less constipation. Safety assessments will include adverse event monitoring, vital signs, laboratory work. starting with 12.5g/h or 25g/h of fentanyl matrix transdermally at the investigator's discretion and flexible dose depending the patient's pain relief for 3 weeks

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed lung cancer, who complain of cancer pain
* Patients who are taking Ultracet, Tramadol, or Codeine (or Codeine combination drug) for cancer pain-relief purposes, but still complain of a pain level of 4 or above on the Numeric Rating Scale (NRS) during the past 24 hours: Ultracet 3 tablets/day, Tramadol 150 mg/day, Codeine 200 mg /day, or Codeine combination less than 3 capsules/day
* Patients who are able to communicate with the investigator about his/her pain
* Patients who use proper contraceptives during the study period if they are women of childbearing potential
* Patients whose life expectancy is 3 months or longer
* Patients who have signed an informed consent form

Exclusion Criteria:

* Patients participating in other clinical trials
* Patients with a history of hypersensitivity to opioid analgesics
* Patients with a history of drug abuse
* Patients who are unable to use a transdermal product due to skin disease
* Patient with a history of CO2 retention (e.g. chronic obstructive pulmonary disease)
* Patients who are receiving radiotherapy or chemotherapy when registering for the study or who plan to receive it during the study
* Patient who are pregnant or are of childbearing potential and not using contraceptives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2006-05; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Patient's satisfaction with pain treatment as measured by 5-point verbal scale | Day 1, 8 and 22

SECONDARY OUTCOMES:
Difference in pain intensity measured by Numeric Rating Scale before and after treatment of the study drug measured | Day 1 (visit 1) and 22 (visit 3)
Detailed reasons for patient's satisfaction with the pain treatment | Day 22 (visit 3)
Patient's and investigator's satisfaction measured by 5-point verbal scale with the study drug | Day 22 (visit 3)
Dose of fentanyl matrix | Day 1 (visit 1), 8 (visit 2) and 22 (visit 3)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd. Clinical Trial, Study Director — Janssen Korea, Ltd.